CLINICAL TRIAL: NCT00116675
Title: A Single-Blind, Dose-Escalating Study to Assess Efficacy and Safety of Resiquimod Gel Applied 3 Times Per Week for 4 Weeks for the Treatment of Common Warts in Pediatric Subjects
Brief Title: Four Week Safety and Efficacy Study With a Topical Gel to Treat Common Warts in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1535-RESI
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2006-06

CONDITIONS: Warts
Keywords: Common Wart(s); Pediatric; Wart(s); Children; 3M Pharmaceuticals; Resiquimod
MeSH Terms: conditions — Warts | interventions — resiquimod

INTERVENTIONS:
Drug: Resiquimod

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness in pediatric subjects of three different strengths of resiquimod gel applied to common wart(s) three times a week for four weeks.

A second purpose is to evaluate the safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of common warts
* Ages between 3 to 11

Exclusion Criteria:

* Other types of wart(s), ie. plantar
* Currently participating in another clinical study
* Chronic viral hepatitis B or C

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84
Dates: Start 2005-03; Study Completion 2006-04

PRIMARY OUTCOMES:
Clearance of treated wart(s)

SECONDARY OUTCOMES:
Partial clearance of treated wart(s)
Wart recurrence

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - University of California - San Francisco, San Francisco, California
  - Longmont Clinic/Longmont Medical Research Network, Longmont, Colorado
  - Mercy Health Research, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rhode Island Hospital - Jane Brown Building, Providence, Rhode Island
  - DermResearch, Inc., Austin, Texas
  - Alpine Pediatrics, Pleasant Grove, Utah
  - Walla Walla Clinic, Walla Walla, Washington
  - Advanced Healthcare, Milwaukee, Wisconsin